CLINICAL TRIAL: NCT04513093
Title: Effect of Abdominal Massage Applied With Ginger and Lavender Oil on Constipation for Elderly Individuals
Brief Title: Aromatherapy Massage Applied on Constipation
Acronym: Aromatherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe Aydınlı (Other)
Responsible Party: Sponsor-Investigator, Ayşe Aydınlı, Dr. Research Asistant, Suleyman Demirel University
Organization: Suleyman Demirel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SuleymanDU Aaydinli
Record Dates: First submitted 2020-08-09; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Constipation
Keywords: Nurse; Elderly; Constipation; Aromatherapy; Abdominal Massage
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): The elderly individuals in the intervention group underwent aromatherapy massage with ginger and lavender oils for a period of five days and 15 minutes on weekdays for four weeks according to the abdominal massage application protocol.
  The "Bristol Stool Scale" and "Constipation Severity Scale" were re-applied to the individuals in the intervention before, during the second week of practice and at the end of practice (fourth week).
  Interventions: Other: Aromatherapy Massage
- Control Group (No Intervention): No application was applied to the individuals in the control group. "Bristol Stool Scale" and "Constipation Severity Scale" were applied to the individuals in the control group at the same time as (at the beginning, second week and fourth week) the intervention group.

INTERVENTIONS:
Other: Aromatherapy Massage — The elderly individuals in the intervention group underwent aromatherapy massage with ginger and lavender oils for a period of five days and 15 minutes on weekdays for four weeks according to the abdominal massage application protocol.
  Arms: İntervention Group

SUMMARY:
Aim: This study was conducted as a randomized controlled experimental study to examine the effect of abdominal massage with ginger and lavender oil on constipation in elderly individuals.

Design: The study was completed with 40 elderly individuals in Kayseri nursing home, including 20 in intervention and 20 in control group who met the criteria for inclusion in the study. In the study, written informed volunteer consent was obtained from the individuals with the approval of the ethics committee and the permission of the institution.

The elderly individuals in the intervention group underwent aromatherapy massage with ginger and lavender oils for a period of five days and 15 minutes on weekdays for four weeks according to the abdominal massage application protocol. No application was made to individuals in the control group.

DETAILED DESCRIPTION:
Aim: This study was conducted as a randomized controlled experimental study to examine the effect of abdominal massage with ginger and lavender oil on constipation in elderly individuals.

Design: The study was completed with 40 elderly individuals in Kayseri nursing home, including 20 in intervention and 20 in control group who met the criteria for inclusion in the study. In the study, written informed volunteer consent was obtained from the individuals with the approval of the ethics committee and the permission of the institution. The data were collected by the researcher using the Questionnaire Form, Bristol Stool Scale, Rome IV Criteria, Constipation Severity Scale and Mini Mental Test.

The elderly individuals in the intervention group underwent aromatherapy massage with ginger and lavender oils for a period of five days and 15 minutes on weekdays for four weeks according to the abdominal massage application protocol. No application was made to individuals in the control group. The "Bristol Stool Scale" and "Constipation Severity Scale" were re-applied to the individuals in the intervention and control group before, during the second week of practice and at the end of practice (fourth week).

ELIGIBILITY:
Inclusion Criteria:

* Elderly individuals with constipation determined by the institution doctor,
* Individuals diagnosed with constipation according to the Roma-criteria,
* Individuals, who achieved a score of 24 and higher on the standardized mini mental test (SMMT),
* Individuals, who do not have lesions disrupting skin integrity in the abdominal region,
* And elderly individuals, who agreed to participate in the study were included.

Exclusion Criteria:

* Individuals diagnosed with irritable bowel syndrome (IBS),
* Individuals who have undergone bowel surgery before,
* Individuals diagnosed with colon cancer,
* Individuals with percutaneous endoscopic gastrostomy,
* Individuals with umbilical hernia
* And individuals allergic to lavender and ginger oil.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
1. Mini Mental Test. | Before the application of massage
  The mini mental test was first developed by Folstein et al. in 1975 to assess cognitive functions. The SMMT consists of five categories, which are orientation, attention and calculation, recall, registration and language. The maximum total score is 30 points. A score higher than 18/19 is considered as good cognitive state for uneducated individuals and a score of 23/34 for educated individuals. The scale was filled out by the researcher before the application by interviewing the elderly participants face to face, who were diagnosed with constipation and agreed to participate in the study.
2. Rome IV Criteria | Before the application of massage
  In this study the diagnosis of constipation was made with the Rome IV criteria. The Rome IV criteria are; straining, lumpy or hard stool, feeling of incomplete emptying, feeling of anorectal obstruction, need for manual intervention, fewer than three defecations per week and rare occurrence of soft stool without laxatives in at least 25% of defecations and insufficient criteria for irritable bowel syndrome. If at least 2 of these symptoms are present and if these symptoms have begun at least 6 months prior or have been lasting for the last three months leads to the diagnosis of constipation.
3. Bristol Stool Scale | in four weeks
  The Bristol Stool Scale was developed by Lewis and Heaton at Bristol University in the United Kingdom. The Bristol Stool Scale provides information about the duration of stool in the colon and its changing physical characteristics during this period and divides the stool types into seven different categories. Type 1 and type 2 describe constipation, type 2, type 4 and type 5 normal stool shapes and type 6 and type 7 diarrhea. The constipation status of the individuals was evaluated with the Bristol Stool Scale three times in total, before the application and in the second and fourth weeks of the application.
4. Constipation Severity Scale | in four weeks
  The Constipation Severity Scale (CSS) consists of 16 questions to determine the frequency of defecation of individuals and the difficulty and pain experienced during defecation. The CSS has three subscales; Obstructive Defecation Subscale (ODSS), Lazy Bowel Subscale (LBSS) and Pain Subscale (PSS). The minimum total score of the CSS is 0 and the maximum score is 73. As the total scale score increases the level of symptoms also increases. In the study, the constipation status of the elderly individuals was evaluated three times in total, before the application and in the second and fourth weeks of the application.

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No